CLINICAL TRIAL: NCT07284043
Title: A Mass Balance Study of [14C] MT1013 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT1013-I-C03
Record Dates: First submitted 2025-11-23; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis Subjects With Secondary Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] MT1013/MT1013 Injection Group (Experimental)
  Interventions: Drug: [14C] MT1013/MT1013 Injection

INTERVENTIONS:
Drug: [14C] MT1013/MT1013 Injection — [14C] MT1013/MT1013 Injection

SUMMARY:
MT1013 is a first-in-class dual-target agonist.This study is being conducted to determine the mass balance and routes of excretion of total radioactivity after the dose of [14C] MT1013.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or postmenopausal female participants, aged 18 years or older, with a confirmed diagnosis of SHPT.
* 2. The BMI is between 18 kg/m2 and 35 kg/m2;
* 3. The subjects must undergo regular maintenance hemodialysis three times a week for at least three months；
* 4. Within 14 days prior to randomization, subjects must have serum calcium levels≥ 8.4 mg/dL;
* 5.Subject capable of understanding written information ,willing to participate in, and provide a written informed consent;

Exclusion Criteria:

* 1. The subjects underwent parathyroidectomy within 6 months prior to screening, or plan to undergo parathyroidectomy or ablation or radiation during the study;
* 2. Gastrointestinal bleeding or peptic ulcer medical history within 6 months prior to screening;
* 3. The subjects had myocardial infarction or had undergone coronary angioplasty or coronary artery bypass grafting within 6 months before screening.
* 4．Subjects with severe uncontrolled hypertension, defined as systolic blood pressure>180 mmHg and/or diastolic blood pressure>110 mmHg;
* 5. History of epileptic seizures or ongoing epilepsy related treatment within 1 year prior to screening;
* 6. History of malignant tumors within the five years prior to screening;
* 7. The subjects received oral cinacalcet or ivocalcet within 7 days before signing the informed consent form, or received Etelcalcetide injection treatment within 4 months.
* 8. Engaged in work that requires long-term exposure to radioactive conditions; Or those who have had significant radioactive exposure or participated in radioactive drug labeling tests within one year prior to screening;
* 9. Participants who may not be able to complete this study for other reasons or who the researchers consider should not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative excretion of radioactivity | Day 1 to Day 91.
Percentage of parent drug and its metabolites in plasma as a percentage of total radioactive exposure (%AUC) | Day 1 to Day 91.

SECONDARY OUTCOMES:
Adverse Events (AEs) | About 13 weeks.
Serious adverse Events (SAEs) | About 13 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital), Jinan, Shandong, China